CLINICAL TRIAL: NCT02683005
Title: Phase I Pharmacokinetic and Safety Trial of Ledipasvir/Sofosbuvir Fixed Dose Combination in Pregnant Women With Chronic Hepatitis C Virus Infection
Brief Title: Study of Hepatitis C Treatment During Pregnancy
Acronym: HIP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Catherine Chappell (Other)
Collaborators: Gilead Sciences (Industry); University of Nebraska (Other)
Responsible Party: Sponsor-Investigator, Catherine Chappell, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO16010091
Record Dates: First submitted 2016-01-25; First posted 2016-02-17 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Hepatitis C; Pregnancy
Keywords: treatment; pharmacokinetics
MeSH Terms: conditions — Hepatitis C | interventions — ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ledipasvir/Sofosbuvir (Experimental): Hepatitis C treatment will be initiated with ledipasvir (400 mg) and sofosbuvir (90mg) fixed dose combination, one pill, once daily for 12 weeks.
  Interventions: Drug: ledipasvir/sofosbuvir

INTERVENTIONS:
Drug: ledipasvir/sofosbuvir — Hepatitis C treatment with ledipasvir and sofosbuvir will be initiated during pregnancy at approximately 24 weeks of gestation.
  Other Names: Harvoni

SUMMARY:
Sofosbuvir and ledipasvir (LDV/SOF) are new directly acting antiviral drugs for the treatment of hepatitis C (HCV) that are highly effective, orally administered, well tolerated and preclinical evaluations in animal models indicate safe administration during pregnancy. This project will evaluate the safety and pharmacokinetics of antenatal LDV/SOF treatment for 12 weeks during the second and third trimester. If proven to be effective, antenatal treatment of HCV with LDV/SOF will prevent maternal HCV-related liver disease, perinatal transmission of HCV, and community transmission of HCV.

DETAILED DESCRIPTION:
There are 3.2 million persons in the United States chronically infected with hepatitis C virus (HCV) with a 1-2.4% prevalence during pregnancy. The recent October 2014 approval of the fixed dose combination, containing the NS5B polymerase inhibitor sofosbuvir (SOF) 90 mg and the NS5A inhibitor ledipasvir (LDV) 400mg, marked a new era of IFN and ribavirin free, directly acting antiviral treatment for HCV. A 12 week treatment course of LDV/SOF resulted in a 99% cure rate when given as a once-a-day oral pill. Based on the animal model data submitted to the FDA, this drug combination was given a pregnancy category B designation, even though there is currently no experience with LDV/SOF in pregnant women.

Pregnancy is a time when women are uniquely motivated to engage in activities which are geared toward improvement of their own health and ensuring the health of their unborn child. As such, pregnant women have frequent prenatal care visits; and health care interventions, such as antiviral therapy and monitoring, can be easily integrated into the existing healthcare infrastructure of prenatal care. The benefits of HCV treatment are numerous, including prevention of severe liver disease, hepatocellular carcinoma, and liver transplantation, as well as improvements physical, emotional and social health. The most recent guidelines by the Infectious Disease Society of America recommend that all HCV-infected persons receive treatment. The antenatal period represents an ideal window of opportunity for treatment of HCV in pregnancy due to increased antenatal health care utilization and prevention of perinatal transmission of HCV to the infant.

Safe administration of drugs in pregnancy may require dose adjustment due to the pregnancy-induced physiologic alternations. Therefore, careful pharmacokinetic (PK) evaluation is a critical first step to ensure safe administration of drugs to both the mother and the developing fetus. This is a single-arm, single-center, open label Phase 1 evaluation of the PK and safety of treating HCV with a 12 week course of LDV/SOF in 15 HCV-infected pregnant women. Therapy will be initiated at approximately 24 weeks of gestation. In this study we will determine: 1) if the PK of the LDV and SOF are similar in pregnancy as compared to those in nonpregnant women, 2) if the viral response to LDV/SOF treatment in pregnancy is similar to that observed in nonpregnant women, and 3) if there are any initial maternal or neonatal safety concerns detected with antenatal LDV/SOF administration compared with HCV-infected historical controls delivered at our institution. From the findings of this study, future studies will seek to optimize the dose, gestational age timing and treatment duration of LDV/SOF during pregnancy. Antenatal HCV treatment will improve maternal health, prevent further HCV transmission in the community and perinatal HCV transmission to the child, and thus enhance the long-term health of two generations.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 through 39 years (inclusive) at Screening
2. Able and willing to provide written informed consent to be screened for and take part in the study procedures
3. Able and willing to provide adequate locator information
4. Chronic HCV, genotype 1, 4, 5, 6 infection, defined as HCV antibody detected at least 6 months prior to Screening and detectable HCV RNA viral load at Screening
5. Desired pregnancy at 23 + 0 to 24 + 6 weeks' gestation at Enrollment with gestational dating confirmed by ultrasound
6. Singleton gestation with no known fetal abnormalities
7. Documented negative Hepatitis B testing for current infection (negative HBsAg test) or previous infection (negative anti-HB Core) performed at the screening visit
8. Negative HIV testing at the screening visit
9. Per participant report at Screening and Enrollment, agrees not to participate in other research studies involving drugs or medical devices for the duration of study participation

Exclusion Criteria:

1. Participant report of any of the following at Screening or Enrollment:

   1. Previous treatment for Hepatitis C virus with an NS5A inhibitor or sofosbuvir
   2. Use of any medications contraindicated with concurrent use of ledipasvir or sofobuvir according to the most current HARVONI package insert
   3. Plans to relocate away from the study site area in the next 1 year and 4 months
   4. Current sexual partner is known to be infected with HIV or Hepatitis B virus
   5. History of cirrhosis documented by previous liver biopsy or liver imaging tests
2. Reports participating in any other research study involving drugs or medical devices within 60 days or less prior to Enrollment
3. Clinically significant and habitual non-therapeutic drug abuse, not including marijuana, as determined by Protocol Chair
4. At Screening or Enrollment, as determined by the Protocol Chair, any significant uncontrolled active or chronic cardiovascular, renal, liver (such as evidence of decompensated cirrhosis by ascites, encephalopathy, or variceal hemorrhage), hematologic, neurologic, gastrointestinal, psychiatric, endocrine, respiratory, immunologic disorder or infectious disease (other than Hepatitis C)
5. Has a high risk of preterm birth defined as a history of spontaneous preterm birth at less than 34 weeks of gestation or a shortened cervical length of less than 20 millimeters
6. Has any of the following laboratory abnormalities at Screening:

   1. Aspartate aminotransferase (AST) or alanine transaminase (ALT) greater than 10 times the upper limited of normal
   2. Hemoglobin less than 9 g/dL
   3. Platelet count less than 90,000 per mm3
   4. International normalized ratio (INR) > 1.5
   5. Creatinine greater than 1.4
   6. Medical history of cirrhosis
7. Has any other condition that, in the opinion of the IoR/designee, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving study objectives.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2020-02-03 (Actual); Study Completion 2020-02-03 (Actual)

PRIMARY OUTCOMES:
Area Under Curve (AUC) Time Frame: predose, 0.5 hr, 1 hr, 2, 3, 4, 5, 8, 12 hrs | 3 gestational age time points during the 12 weeks of treatment: 1) Between 25 + 0 and 26 + 5; 2) Between 29 + 0 and 30 + 6; 3) 33 + 0 and 34 + 6 weeks' gestation
  Systemic exposure both LDV and SOF (SOF and inactive metabolite GS-331007) will be assessed at 3 gestational age time points: 1) Late second trimester between 25 + 0 and 26 + 5 weeks' gestation (after at least 10 days of therapy); 2) Early third trimester between 29 + 0 and 30 + 6 weeks' gestation; 3) Late third trimester between 33 + 0 and 34 + 6 weeks' gestation

SECONDARY OUTCOMES:
Sustained viral response at 12 weeks post treatment (SVR 12) | -HCV RNA viral load will be assessed at 12 weeks after completion of LDV/SOF treatment
  An undetectable HCV viral load is considered an SVR 12.
Number of Maternal Adverse Events | -From enrollment to 12 weeks after treatment completion
  Adverse events, including pregnancy and delivery outcomes will be collected prospectively . -
Number of Participants With Abnormal Laboratory Values | -From enrollment to 12 weeks after treatment completion
  Safety laboratories will be sent 4-6 weeks after the initiation of treatment and will include CBC, chemistries, liver function tests, creatinine kinase, lipase, and coagulation studies.
Major Malformations of the Neonate | From birth until 1 year of life
  Major malformations, defined as structural abnormalities with surgical, medical, or cosmetic importance
Length | From birth until 1 year of life
  Length in centimeters will be collected at birth, 1 month, 6 months, and 12 months.
Weight | From birth until 1 year of life
  Weight in kilograms will be collected at birth, 1 month, 6 months, and 12 months.
Head circumference | From birth until 1 year of life
  Head circumference (centimeters) will be collected at birth, 1 month, 6 months and 12 months.
Perninatal Hepatitis C Transmission | From birth until 1 year of life
  Perinatal HCV transmission assessed by presence of hepatitis C virus RNA from infant blood sampling at one month, six months and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine A Chappell, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee Womens Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chappell CA, Scarsi KK, Kirby BJ, Suri V, Gaggar A, Bogen DL, Macio IS, Meyn LA, Bunge KE, Krans EE, Hillier SL. Ledipasvir plus sofosbuvir in pregnant women with hepatitis C virus infection: a phase 1 pharmacokinetic study. Lancet Microbe. 2020 Sep;1(5):e200-e208. doi: 10.1016/S2666-5247(20)30062-8. Epub 2020 Jul 27. PMID 32939459